CLINICAL TRIAL: NCT03993340
Title: Rescue Stenting for Failed Endovascular Thrombectomy in Acute Ischemic Stroke (ReSET)
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-1148
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Acute Ischemic Stroke; Intracranial Artery Occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Rescue stenting group
  Interventions: Device: Rescue stenting

INTERVENTIONS:
Device: Rescue stenting — The subjects will receive endovascular treatment for acute stroke according to standard clinical practice. Specifically, modern endovascular thrombectomy using a stent retriever, contact aspiration thrombectomy, or both are allowed. The number of thrombectomy attempts is at the operator's discretion. After failure of standard thrombectomy procedure, rescue stenting with Solitaire will be done. Additional balloon angioplasty, glycoprotein IIb/IIIa inhibitor (GPI), or thrombolytic infusions are optional and at the operator's discretion. After successful recanalization with rescue stenting, intravenous maintenance of GPI at least for a 12 hours and then changed to oral antiplatelet are recommended.

SUMMARY:
This study is a prospective, open-label, multi-center, registry study, designed to show that rescue stenting is safe and effective for emergency large vessel occlusion (ELVO) patients who have mechanical thrombectomy failure. Participants with ELVO will initially underwent mechanical thrombectomy usig stent retriever, contact aspiration or both. After failure of mechanical thrombectomy, rescue stenting will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects experiencing acute ischemic stroke due to large vessel occlusion (intracranial internal carotid artery and middle cerebral artery M1 segment)
* 2. Age 19 or greater
* 3. mRS before qualifying stroke, 0 or 1
* 4. Baseline NIHSS score 4 or more
* 5. CT ASPECTS > 6 or MR ASPECTS > 5
* 6. Good collateral statues on CT angiogram (collateral grade by Calgary group, 4 or 5) or corresponding to DEFUSE 3 or DAWN trial on perfusion imaging.
* 7. Onset (last-seen-well) time to femoral puncture time < 24 hours
* 8. Failure of mechanical thrombectomy with stent retriever, contact aspiration or both
* 9. Subjects who received rescue stenting after failure of mechanical thrombectomy
* 10. Anticipated life expectancy of at least 12 months
* 11. Signed informed consent for study enrollment

Exclusion Criteria:

* 1. Any contraindication to antiplatelet medication
* 2. Multiple simultaneous large vessel occlusions
* 3. Pregnancy
* 4. Severe contrast allergy or absolute contraindication to iodinated contrast agent
* 5. Patient has a severe or fatal combined illness that will prevent improvement of follow-up or will render the procedure unlikely to benefit the patient.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with emergent large vessel occlusion and who have not achieved successful recanalization (defined by mTICI, 2b or 3) by mechanical thrombectomy using stent retriever or aspiration thrombectomy.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
modified Rankin scale | 3 months
  The rate of good functional outcome defined by modified Rankin Scale score, 0 - 2

SECONDARY OUTCOMES:
Patency of the target artery | 1 day to 28 days
  The rate of patency of the treated artery at follow-up vascular imaging (magnetic resonance angiography, computed tomography angiography, or catheter angiography)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital Stroke Center, Yonsei University College of Medicine, Seoul, Yeonsei-ro Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No